CLINICAL TRIAL: NCT04212962
Title: Evaluation of the Multisite Replication of the Transitional Care Model
Brief Title: Transitional Care Model Evaluation 2020
Acronym: TCM2020
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Mathematica Policy Research, Inc. (Other)
Collaborators: University of Pennsylvania (Other); Arnold Ventures (Unknown); Veterans Health Administration--St. Louis and Cleveland (Unknown); Trinity Health System (Industry); Providence St. Joseph Health-Swedish Health Services (Swedish) (Unknown); University of California, San Francisco (Other)
Responsible Party: Principal Investigator, Randy Brown, Principal investigator, Mathematica Policy Research, Inc.
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: MathematicaPR
Record Dates: First submitted 2019-12-24; First posted 2019-12-30 (Actual); Last update posted 2023-03-16 (Actual); Status verified 2023-03

CONDITIONS: CHF - Congestive Heart Failure; COPD; Pneumonia
MeSH Terms: conditions — Heart Failure; Pulmonary Disease, Chronic Obstructive; Pneumonia

STUDY DESIGN:
Intervention Model Description: Advance practice registered nurses provide care management and education to intervention group patients prior to discharge and during the 90 days after transitioning to home.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment group (Experimental): The treatment group receives the TCM intervention while in the hospital and during the first 90 days after returning to the community.
  Interventions: Behavioral: Transitional care model (TCM)
- Control group (Experimental): The control group receives usual discharge planning and post-discharge care.
  Interventions: Behavioral: Usual care

INTERVENTIONS:
Behavioral: Transitional care model (TCM) — Patient education about post-discharge self-care and medications, arrangement of needed social services, coordination of information from medical providers interacting with patient
  Arms: Treatment group
Behavioral: Usual care — usual hospital discharge and post-discharge care
  Arms: Control group

SUMMARY:
The study is a randomized controlled trial to estimate the effects of the transitional care model (TCM) on hospital admissions and patients' experience during the year following the patient's qualifying discharge. The University of Pennsylvania, where TCM was developed, will be the coordinating center for the implementation. The study will be conducted in three large health systems spread throughout the U.S., drawing patients from seven hospitals in those systems. Eligible patients are older adults (age 65 and older) admitted to a participating hospital with symptoms of heart failure (HF), chronic obstructive pulmonary disease (COPD), or pneumonia (PNA). The evaluation will be conducted by Mathematica.

DETAILED DESCRIPTION:
The Transitional Care Model (TCM) is an advanced practice registered nurse (APRN) led, team-based, care management strategy designed to improve the care and outcomes of high-risk older adults transitioning from hospital to home. Eligible patients who agree to participate in the study will be randomly assigned to either the intervention group, which receives the TCM intervention, or the control group, which receives usual care (standard hospital discharge planning and post-hospital follow up services). The target sample size for the study is close to 1000, evenly divided into intervention and control groups, with 250 to 270 patients derived from each of UCSF and Trinity health systems, and another 450 recruited from the two VHA hospitals combined. Data will be collected at intake, prior to randomization, by enrollment coordinators at each of the participating hospitals. Followup data will be collected in a survey of patients conducted 90 days after discharge, and from claims data obtained from Medicare, Medicare Advantage plans, and the VHA.

ELIGIBILITY:
Inclusion Criteria:

* Age 65 years and older
* Admitted from home with Pneumonia OR with a history of HF or COPD with symptoms of HF or COPD exacerbation or whose symptoms suggest a new HF or COPD diagnosis
* English and non-English speaking, able to respond to questions
* Reachable by telephone after discharge
* Resides within the geographic service area
* Consent to participation

Exclusion Criteria:

* Enrolled in Medicare's Hospice or End-Stage Renal Disease programs
* Presence of active and untreated psychiatric conditions (ICD10: F10-F29)
* Long-term care resident
* Undergoing active cancer treatment
* Currently enrolled in another RCT

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 962 (Actual)
Dates: Start 2020-07-07 (Actual); Primary Completion 2024-07 (Estimated); Study Completion 2025-02 (Estimated)

PRIMARY OUTCOMES:
Number of hospital admissions | 12 months
  number of times admitted to the hospital during 12 months after initial discharge
Costs | 12 months
  Costs of medical care paid for by Medicare, Medicare Advantage plan, or Veterans Health Administration

SECONDARY OUTCOMES:
30-day readmission | 30 days
  whether readmitted to a hospital during the 30 days after initial discharge
emergency department visits | 12 months
  number of times treated in an emergency department after initial discharge
Mortality | 12 months after initial discharge
  whether died after initial discharge
Edmonton Symptom Assessment Scale | 90 days after initial discharge
  measures post-hospital symptoms, range 0-100, high score is bad
Patient-Reported Outcomes Measurement Information System Physical Functioning (SF10a) | 90 days after initial discharge
  functional status, range 10-50, high score is good
Patient Health Questionnaire for Depression and Anxiety (PHQ-4) | 90 days after initial discharge
  index of depression and anxiety, range 0-12, high score is bad

OTHER OUTCOMES:
Skilled nursing facility days | 12 months after initial discharge
  Number of days spent in a skilled nursing facility
Home Health | 12 months after initial discharge
  number of home health visits
length of time to death or hospital admission | 12 months after initial discharge
  number of days between initial discharge and either death or readmission to hospital
hospice | 12 months after initial discharge
  whether admitted to hospice care

CONTACTS AND LOCATIONS:
Overall Officials: Arkadipta Ghosh, PhD, Study Director — Mathematica Policy Research, Inc.; Randall S Brown, PhD, Principal Investigator — Mathematica Policy Research, Inc.
Locations (1):
- Mathematica Policy Research, Princeton, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Naylor MD, Aiken LH, Kurtzman ET, Olds DM, Hirschman KB. The care span: The importance of transitional care in achieving health reform. Health Aff (Millwood). 2011 Apr;30(4):746-54. doi: 10.1377/hlthaff.2011.0041. PMID 21471497
- [Background] Naylor MD, Brooten D, Campbell R, Jacobsen BS, Mezey MD, Pauly MV, Schwartz JS. Comprehensive discharge planning and home follow-up of hospitalized elders: a randomized clinical trial. JAMA. 1999 Feb 17;281(7):613-20. doi: 10.1001/jama.281.7.613. PMID 10029122
- [Background] Naylor MD, Brooten DA, Campbell RL, Maislin G, McCauley KM, Schwartz JS. Transitional care of older adults hospitalized with heart failure: a randomized, controlled trial. J Am Geriatr Soc. 2004 May;52(5):675-84. doi: 10.1111/j.1532-5415.2004.52202.x. PMID 15086645
- [Derived] McHugh M, Hirschman KB, Toles MP, Ahrens M, Morgan B, Osokpo O, Shaid EC, McCauley K, Hanlon AL, Pauly MV, Naylor MD. Implementing the MIRROR-TCM Randomised Control Trial During the COVID-19 Pandemic: A Mixed-Methods Evaluation. J Adv Nurs. 2025 Nov;81(11):7835-7854. doi: 10.1111/jan.16594. Epub 2024 Nov 25. PMID 39582355
- [Derived] Naylor MD, Hirschman KB, Morgan B, McHugh M, Hanlon AL, Ahrens M, McCauley K, Shaid EC, Pauly MV. The study protocol to evaluate implementation of the transitional care model in four U.S. healthcare systems during the Covid-19 pandemic. Arch Gerontol Geriatr. 2023 May;108:104944. doi: 10.1016/j.archger.2023.104944. Epub 2023 Jan 25. PMID 36709563